CLINICAL TRIAL: NCT02042651
Title: Low Intensity Extracorporeal Shockwave Therapy Against Chronic Pelvic Pain: a Randomized and Sham Controled Study
Brief Title: A Sham Controlled Study of the Effects of Ultrasonic Shockwaves as a Treatment for Chronic Pelvic Pain
Acronym: CPPESWT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study stopped because of insuficient number of comparable patients available.
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Anders Frey, Junior researcher, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H-3-2013-178; HEH-2013-33 (Other: The danish dataprotection agency)
Record Dates: First submitted 2014-01-10; First posted 2014-01-23 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Pelvic Pain
Keywords: ESWT; Chronic pelvic pain; randomized; sham controlled

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low intensity extracorporeal shockwave therapy (Experimental): Active treatment with low intensity extracorporeal shockwave therapy applied to the perineum.
  Interventions: Device: Low intensity extracorporeal shockwave therapy
- Sham low intensity extracorporeal shockwave therapy (Sham Comparator): Sham treatment with low intensity extracorporeal shockwave therapy applied to the perineum.
  Interventions: Device: Sham low intensity extracorporeal shockwave therapy

INTERVENTIONS:
Device: Low intensity extracorporeal shockwave therapy — Shockwaves will be applied to the perineum a total of 6 times once per week. The energy level applied will range between 0.25 and 0.40 mJ/mm2 with a frequency of 3 Hz for a total of 3000 shockwaves per treatment session
  Other Names: Storz Duolith® SD1 T-TOP, CE 1275
  Arms: Low intensity extracorporeal shockwave therapy
Device: Sham low intensity extracorporeal shockwave therapy — Shockwaves will be applied to the perineum a total of 6 times once per week. The shockwaves will be blocked by a medium on the handheld applicator.
  Other Names: Storz Duolith® SD1 T-TOP, CE 1275
  Arms: Sham low intensity extracorporeal shockwave therapy

SUMMARY:
Introduction:

Chronic pelvic pain with unknown pathology is a condition that affects both men and women. the condition is defined as pelvic pain lasting for a minimum of 6 months without any known etiology eg. cancer, infection or inherent anatomical abnormalities. Low intensity extracorporeal shockwave therapy (LIESWT) enables the practitioner to deliver a small amount of energy approximately 5 cm under the skin of the patient without damaging the skin. This have been shown to increase blood flow and accelerate healing which could also be beneficial in chronic pelvic pain patients.The purpose of this study is to investigate the effects of LIESWT on chronic pelvic pain.

Methods:

All patients will be treated at the Birthe Bonde clinic, in Copenhagen, Denmark.

The investigators anticipate to include 100 chronic pelvic pain patients in the study.

included patients will be randomized into two groups: active treatment or sham treatment.

All patients will be required to provide a urine sample and a semen sample prior to final inclusion. Samples will be analyzed for microbial growth. Furthermore, patients will undergo a digital rectal exploration and finally all patients is required to provide an informed consent in order to be included in the study.

A Storz Doulith SD1 T-Top (CE1275) will be used to generate shockwaves. Patients will receive the treatment once a week until their symptoms have seized or for a maximum of 6 times. Each treatment consists of 3000 shockwaves applied to the perineum with a energy density of 0.25-0.40 millijoule(mJ)/mm2 and a frequency of 3 hz.

Participants will fill out a questionnaire one week before the treatment, one week, four weeks, and twelve weeks after the last treatment.

Possible gains from this study:

The investigators hope to provide further evidence for this treatment and consequently be able to offer the treatment as an alternative to the very limited array of treatments existing for this group of patients today.

Ethics, funding, and publication:

The study is performed in compliance with the Helsinki declaration. External funding have been applied for but not yet received. Participants will be informed of sources of external funding. The result of the study will be published as soon as possible, preferably in a peer-reviewed international journal.

ELIGIBILITY:
Inclusion Criteria:

* pelvic pain with a duration of more than 6 months
* be able to read and understand the study information

Exclusion Criteria:

* known etiology for pelvic pain eg. cancer, infection, inherent abnormalities.
* diagnosed with hemophilia
* receiving anti thrombotic therapy other than hearth magnyl
* diagnosed with thrombocytosis
* active cancer
* treated with IV glucocorticoids within the last 6 months
* disease in the rectal area
* abnormal digital rectal exploration
* bacteriospermia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Change in NIH-Chronic Prostatitis Symptom Index | Change from baseline to twelve weeks after final treatment
  A questionnaire designed to provide symptom scores for patients with chronic prostatitis. The index provides scores on pain, urinary symptoms, and quality of life.

SECONDARY OUTCOMES:
Change in The International Index of Erectile Function 5 | Change from baseline to twelve weeks after final treatment
  Questionnaire designed to evaluate erectile capabilities. The questionnaire provides a score between 5 and 25.
Change in The International prostate symptom score | Change from baseline to twelve weeks after final treatment
  A questionnaire designed to provide information on lower urinary tract symptoms and their impact on quality of life. scores range from 0 to 35.
Global satisfaction score | Twelve weeks after final treatment
  One question designed to estimate treatment satisfaction on a four point Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Anders U Frey, Bach. Med., Principal Investigator — Urological Research Unit, Herlev Hospital
Locations (1):
- Birthe bonde klinikken, Copenhagen E, Copenhagen, Denmark